CLINICAL TRIAL: NCT02041442
Title: Pilot of Electrophysiologic Mapping of the Urinary Bladder
Brief Title: Electrophysiologic Mapping of the Bladder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study to be redesigned based on initial results
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E-13-529
Record Dates: First submitted 2014-01-16; First posted 2014-01-22 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Electrical Evaluation of Urinary Bladder
Keywords: overactive bladder; cystoscopy
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): Electrical mapping of the urinary bladder
  Interventions: Procedure: Electrical mapping of the urinary bladder

INTERVENTIONS:
Procedure: Electrical mapping of the urinary bladder

SUMMARY:
The hypothesis is that the intrinsic electrical activity of the urinary bladder in response to filling is detectable and can be mapped. This is a pilot study to evaluate the feasibility of using cardiac electrical mapping catheters to measure bladder voltage in patients at the time of routine urodynamic and cystoscopic evaluation.

DETAILED DESCRIPTION:
This pilot study is looking at the possibility of adapting some of the tools and techniques used by cardiac electrophysiologists (doctors specializing in the electrical activity of the heart) to help diagnose and treat Overactive Bladder. The rationale for this approach is based on the similarities of the two organs. In simple terms, the heart and bladder are both hollow muscular organs that expand and contract to hold and move fluid.

In an electrophysiology study looking at cardiac (heart) arrhythmia (irregular heartbeat), the cardiologist places one or more electrode catheters (thin hollow tube with an electrical conductor on the end) through a vein or artery in the leg or arm to contact heart tissue. By recording the electrical activity at multiple sites of the heart, the catheter allows for mapping of the electrical activity and the arrhythmia mechanism.

In this study, investigators will use the same electrode catheter to contact bladder tissue, introduce a low frequency current, and map the electrical activity of the bladder. A sterile cardiac electrical mapping catheter will be used to make contact with the walls of the bladder and introduce a low frequency current starting with the trigone and then the four quadrants of the dome. Electrical activity will be recorded for each volumetric milestone at each location. It is hoped that the information from this electrophysiological testing of the bladder may eventually lead to treatment of areas of electrical abnormality of interest. No actual treatment of the bladder will be done as part of this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a female > = 18 years old.
* Subject is willing and able to provide informed consent.
* Subject has subjective and objective evidence for urinary urgency (with or without incontinence), stress incontinence, or mixed incontinence (with features of both urgency and stress).
* Subject requires urodynamic/cystoscopic studies to complete their workup.

Exclusion Criteria:

* Active urinary tract infection
* Pregnant women
* Patients on anticholinergic medicine for overactive bladder
* Patients with history of intravesical botulinum toxin injections
* Patients with a sacral neuromodulator implant
* Patients with a history of urinary tract malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in electrical activity | 3 months
  goal of this pilot study is to determine whether electrical activity can be recorded from different areas of the bladder using cardiac surface electrodes

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vardy, MD, Principal Investigator — Englewood Hospital and Medical Center
Locations (1):
- Englewood Hospital and Medical Center, Englewood, New Jersey, United States